CLINICAL TRIAL: NCT02844712
Title: Negative Predictive Value of Drug Provocation Tests to Beta-lactams
Acronym: NPVDPT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of the period of inclusion, NSN not achieved
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 9394
Record Dates: First submitted 2016-07-15; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Drug Hypersensitivity
Keywords: Drug hypersensitivity; Betalactam; Drug provocation test
MeSH Terms: conditions — Drug Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Evaluation of reexposure to a negatively tested betalactam (Other)
  Interventions: Other: Evaluation of reexposure to a negatively tested betalactam

INTERVENTIONS:
Other: Evaluation of reexposure to a negatively tested betalactam

SUMMARY:
Patients with a complete drug allergy work-up to betalactam antibiotics were contacted (by mail) and asked to answer a questionnaire regarding the tolerance upon readministration of a negatively tested beta-lactam.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients with at least 5 years at the time of consultation for allergy suspected allergy to beta-lactam antibiotics in the University Hospital of Montpellier and with a negative provocation test to a betalactam
* The patient or the patient's legal representatives are not their opposition to participate in this study
* The patient must be affiliated or beneficiary in a health insurance system

Exclusion Criteria:

* The patient is exclusion period determined by a previous study
* The patient is under judicial protection, guardianship or curatorship
* The patient or the patient's legal representatives do not read fluently the French language

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2014-12; Primary Completion 2016-05 (Actual); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Negative predictive value of drug provocation tests to betalactams | one day

SECONDARY OUTCOMES:
The types of reactions upon reexposure to a negatively tested betalactam | one day

CONTACTS AND LOCATIONS:
Locations (1):
- Allergy Unit, Arnaud de Villeneuve Hospital, University Hospital of Montpellier, Montpellier, France